CLINICAL TRIAL: NCT02505971
Title: Nadolol Versus Propranolol in Children With Infantile Hemangiomas: a Randomized, Controlled, Double-blinded Trial
Brief Title: Nadolol Versus Propranolol in Children With Infantile Hemangiomas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Elena Pope, Section Head, Dermatology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000048673
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Infantile Hemangioma
Keywords: hemangioma, propranolol, nadolol
MeSH Terms: conditions — Hemangioma, Capillary; Hemangioma | interventions — Nadolol; Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nadolol group (Active Comparator): 40 study participants will take Nadolol (oral liquid suspension)
  Interventions: Drug: Nadolol
- Propranolol group (Active Comparator): 40 study paticipants will take Propranolol (oral liquid suspension)
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Nadolol — Patients will be administered twice-daily doses of medication as follows: since Day 0- 0.5 mg/kg/day ; since Day 7-1.0 mg/kg/day and since Day 14- 1.5 mg/kg/day. In all subsequent visits the dosage will be adjusted based on the current weight rather than the baseline weight to maintain 1.5 mg/kg/day. Or the dose may be escalated (by 0.5 mg/kg/day at any following study visit) up to 3 mg/kg/day based on the clinical response to maintain the dose that led to at least 75% reduction in the hemangioma size until Week 24, when unblinding happen. At Week 24 paticipants can start weaning by 10% per week or continue with the last dose, depending on the investigator's decision.
  S/he will be monitored until Week 52.
  Other Names: N/A (any brand )
  Arms: Nadolol group
Drug: Propranolol — Patients will be administered twice-daily doses of medication as follows: since Day 0- 0.5 mg/kg/day ; since Day 7-1.0 mg/kg/day and since Day 14- 1.5 mg/kg/day.
  In all subsequent visits the dosage will be adjusted based on the current weight rather than the baseline weight to maintain 1.5 mg/kg/day. Or the dose may be increased by investigator, based on clinical response by 0.5 mg/kg/day at any study visit (up to 3 mg/kg/day divided twice a day) to maintain the dose that lead to at least 75% reduction in the hemangioma size until Week 24, when unblinding happen. At Week 24 paticipants can start weaning by 10% per week or continue with the last dose, depending on the investigator's decision.
  S/he will be monitored until Week 52.
  Other Names: N/A (any brand)
  Arms: Propranolol group

SUMMARY:
The purpose of this study is to assess the efficacy and safety of oral propranolol versus nadolol in patients with Infantile Hemangiomas (IH) in a randomized, controlled, double-blinded study.

DETAILED DESCRIPTION:
The study objective is to compare the efficacy and safety of oral propranolol in comparison with oral nadolol in patients with IH. Patients will be randomly assigned to either propranolol or dose equivalent nadolol. The duration of the study will be 24 weeks, however, patient will be monitored for up to 1 year post study enrolment. Both efficacy and safety will be closely monitored and captured.

ELIGIBILITY:
Inclusion Criteria:

* 1-6 months corrected age
* Written parental informed consent
* At least one of the following:

  * Size: hemangioma >1.5 cm on the face or >3 cm on other body parts
  * Causing or with potential for functional impairment (e.g. amblyogenic IH, ulcerated hemangioma)
  * Causing or with potential for cosmetic disfigurement (e.g. nasal tip, glabella location)

Exclusion Criteria:

* Contraindications to beta-blockers

  * Hypotension
  * Bradycardia
  * Hypoglycemia
  * Cardiac disease associated with decreased ejection fraction and/or > second degree heart block
  * Bronchospasm (including bronchial asthma)
  * Allergic rhinitis
* Corrected gestational age less than 1 month at screening
* Patients with PHACES cerebral arteriopathy at risk of stroke
* Patients and/or breastfeeding mothers receiving treatment with anti-arrhythmic agents, calcium channel blockers, ACE inhibitors, inotropic agents, vasodilators, hypoglycemic agents, neuroleptics, antiacids, benzodiazepines, thyroxine, warfarin
* Patients treated with an oral beta-blocker or other agent (e.g. systemic steroids, vincristine) within 2 weeks from randomization
* Patients treated with topical timolol within 1 week from randomization
* Vascular tumors other than infantile hemangioma (e.g. pyogenic granuloma, hemangioendothelioma)

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2015-09; Primary Completion 2020-04 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The change in the bulk (size/extent) and color of the infantile hemangioma (IH)at Week 24 compared to baseline using Visual Analog Scale (VAS). | 24 weeks
  A 100 mm visual analog scale (VAS) will be used to quantify changes in the visible bulk (size/extent) and color of the lesion by comparing clinical photographs at 24 weeks versus baseline

SECONDARY OUTCOMES:
Percent change in IH bulk using VAS at 4, 12, 52 weeks | 4, 12, 52 weeks
  A 100 mm visual analog scale (VAS) will be used to quantify changes in the visible bulk (size/extent) of the lesion by comparing clinical photographs at weeks 4, 12, and 52 versus baseline
Time and dose to reach the 50%, 75% and 100% tumor shrinkage | 52 weeks
  Time frame since the baseline and study medication dose, when patient's IH decreased in size by 50%, 75% and 100%.
Inter-rater reliability of the VAS scores | 52 weeks
  Two raters will assess the changes in IH for each study patient ( each visit). We will compare these results to assess inter-rater reliability.
Percentage of patients achieving functional correction at Week 4, 12, 24, 52 | 4,12,24,52 weeks
  Percentage of patients achieving functional correction at Week 4, 12, 24, 52
Percent change in the volumetric changes of hemangioma | 24 and 52 weeks
  [(Length + Width)/2]3 X 0.07
Percentage of patients with residual changes (telangiectasias, discoloration, fibro-fatty changes, anetoderma) | 52 weeks
  Percentage of patients with residual changes
Frequency of observed and reported adverse events | 52 weeks
  Frequency of observed and reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Elena Pope, MD, MSc, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Pope E, Lara-Corrales I, Sibbald C, Liy-Wong C, Kanigsberg N, Drolet B, Ma J. Noninferiority and Safety of Nadolol vs Propranolol in Infants With Infantile Hemangioma: A Randomized Clinical Trial. JAMA Pediatr. 2022 Jan 1;176(1):34-41. doi: 10.1001/jamapediatrics.2021.4565. PMID 34747977